CLINICAL TRIAL: NCT06496919
Title: A Multicenter Real-world Research on the Prevention and Treatment of Peritoneal Metastasis and Malignant Ascites by Intraperitoneal Infusion of rmhTNF in Gastric and Colorectal Malignant Tumors
Brief Title: A Real-world Research on the Prevention and Treatment of Peritoneal Metastasis and Malignant Ascites by Intraperitoneal Infusion of rmhTNF in Gastric and Colorectal Malignant Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Bin Xiong, MD, Chief Physician, Wuhan University
Other Study IDs: PM-GCCC-TNF
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer
Keywords: rmhTNF, gastric cancer, colorectal cancer, peritoneal metastasis, intraperitoneal infusion chemotherapy
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric malignant tumor queue
  Interventions: Drug: Recombinant Mutant Human Tumor Necrosis Factor
- Colorectal Malignant Tumor Queue
  Interventions: Drug: Recombinant Mutant Human Tumor Necrosis Factor

INTERVENTIONS:
Drug: Recombinant Mutant Human Tumor Necrosis Factor — The patients who received rmhTNF intraperitoneal perfusion (intraperitoneal surgical field flushing perfusion or intraperitoneal thermal perfusion chemotherapy)

SUMMARY:
Peritoneal metastasis is the main factor leading to poor prognosis in patients with gastric cancer or colorectal cancer. Although current systemic treatment regimens can prolong the time to peritoneal metastasis, the long-term survival rate is still poor. This is mainly due to the presence of the peritoneal plasma barrier, which limits the penetration of anti-tumor drugs and thus restricts the efficacy. In contrast, the use of intraperitoneal infusion chemotherapy allows anti-tumor drugs to directly reach the abdominal cavity, exposing metastatic nodules to high concentrations of drugs, and has a significant therapeutic effect on peritoneal metastases, resulting in better therapeutic effects Tumor necrosis factor (TNF) is a small molecule protein secreted by macrophages. There are two types of TNF - α: α and ß. TNF - α is produced by activated monocytes and macrophages, also known as cachectin. TNF - α is produced by activated lymphocytes, also known as lymphotoxins, and the two have similar activity. Previous studies have shown that rmhTNF is safe for intraoperative perfusion in gastrointestinal tumors.

In this real-world study, we will observe the safety and effectiveness of rmhTNF intraperitoneal perfusion in actual clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* 1. The initial pathological diagnosis is gastric adenocarcinoma and colorectal adenocarcinoma, with clinical stage progression or advanced stage (cII-IV stage).

  2. Patients with recurrent/metastatic gastric adenocarcinoma and colorectal cancer.

  3. Age range from 18 to 80 years old; 4. Male or non pregnant or lactating female; 5. The bone marrow reserve function is good, and the blood routine meets the following conditions: white blood cell count ≥ 3.5 × 109/L, neutrophils ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, hemoglobin ≥ 90 g/L; 6. The organ function is good, and the biochemical examination meets the following conditions: ALT ≤ 2.5 x Upper Limit of Normal (ULN), AST ≤ 2.5 x ULN, serum total bilirubin ≤ 1.5 x ULN, and blood creatinine ≤ 1.5 x ULN; 7. Functional status: 0-1 (ECOG); 8. preoperative ASA grading I-III; 9. Informed consent form has been signed for clinical treatment.

Exclusion Criteria:

* 1. Individuals who are allergic to TNF, biological products, or penicillin; 2. Those who do not meet the inclusion criteria during pregnancy or lactation; 3. Other situations where the researcher believes that patients are not suitable to participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The initial pathological diagnosis is gastric adenocarcinoma and colorectal adenocarcinoma, with clinical stage progression or advanced stage (cII-IV stage).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) | after radical surgery for 1-3 years
  Postoperative peritoneal implantation metastasis rate of gastric and colorectal adenocarcinoma
Progression-Free Survival （PFS） | after radical surgery for 3 years
  Survival without peritoneal implant metastasis after radical surgery for gastric and colorectal adenocarcinoma
Objective Response Rate | after radical surgery for 3 years
  Objective Response Rate of peritoneal metastasis in gastric and colorectal adenocarcinoma
Disease Control Rate | 4 weeks after administration
  Disease Control Ratel rate of malignant ascites in gastric and colorectal adenocarcinoma

SECONDARY OUTCOMES:
Overall Survival（OS） | after radical surgery for 3 years
  Time from the first study treatment until death from any cause
Regional recurrence rate | after radical surgery for 3 years
  Regional recurrence rate after radical surgery for gastric and colorectal adenocarcinoma (Local recurrence after radical surgery for gastric cancer refers to the recurrence of the duodenal stump, tumor bed, and residual stomach after anastomosis, Bi II style anastomosis, as well as the recurrence of regional lymph nodes)
Adverse events | 24 hours after administration
  The safety of rmhTNF intraperitoneal perfusion therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bin Xiong, Doctor, Principal Investigator — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China